CLINICAL TRIAL: NCT03513367
Title: The Validation Process for Confirmation of the French Version of the Pediatric Quality of Life Inventory (PedsQLTM) 3.0 Duchenne Muscular Dystrophy Module.
Brief Title: The Validation Process for Confirmation of the French Version of the Pediatric Quality of Life Inventory :PedsQLTM.
Acronym: ValPedsQLDMD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/18/0119; 2018-A00895-50 (Other: ID-RCB)
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy,; Pediatric Quality of Life Inventory; disability paradox
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Boys with Muscular Duchenne Dystrophy: 105 boys with Muscular Duchenne Dystrophy (DMD) distributed as follows: 35 patients with Duchenne muscular dystrophy by age category, 8-12 years old and 13-18 years old.
  Children will complete the questionnaire of Duchenne Muscular Dystrophy of the PedsQL ™ 3.0 scale regardless of his parents
  Interventions: Other: Duchenne Muscular Dystrophy of the PedsQL ™ 3.0 scale; Other: The following data of motor function
- Parents of boys with Muscular Duchenne Dystrophy: 105 parents of boys with Muscular Duchenne Dystrophy For the 5-7 age group, only parents answer the questionnaire but medical data are collected : 35 by age category (5-7; 8-12; 13-18) Parents will complete the questionnaire of Duchenne Muscular Dystrophy of the PedsQL ™ 3.0 scale regardless of their children
  Interventions: Other: Duchenne Muscular Dystrophy of the PedsQL ™ 3.0 scale

INTERVENTIONS:
Other: Duchenne Muscular Dystrophy of the PedsQL ™ 3.0 scale — Scaling in multidisciplinary consultations in the form of a self-administered questionnaire with the help of a third party (psychologist). The child and his / her parent complete the questionnaire independently. The result of the questionnaire will then be scored.
  To validate the French translation of the pediatric module of Duchenne Muscular Dystrophy of the PedsQL ™ 3.0 scale. The validation process is confirmatory, the scale being widely used in English. The scale will measure the quality of life of the child using two independent assessments : children and their parents.
Other: The following data of motor function — In parallel, the following data are collected on the day of the consultation: assessment of motor function (MFM, use of a wheelchair, age of loss of walking); assessment of respiratory function (EFR, FVC, respiratory assistance, type of respiratory aid); evaluation of cardiac function (FE); assessment of nutritional status (weight, height, BMI, nutritional support by gastrostomy), school status; ongoing drug treatments (corticosteroids, IEC).
  Groups: Boys with Muscular Duchenne Dystrophy

SUMMARY:
There isn't specific Health related quality of life measure for children with DMD in French. The aim of this study is to validate the French version of the Pediatric Quality of Life Inventory 3.0 Duchenne Muscular Dystrophy module with a multicentric study. The investigators will evaluate the following psychometric properties : convergent validity, internal validity, inter-rater reliability. The investigators would like to be able to use this scientific tool in future clinical trials.

DETAILED DESCRIPTION:
The Duchenne Muscular Dystrophy, the commonest form of dystrophy, is an X-linked, recessive neuromuscular disease, in which there is an absence of the protein dystrophin. This chronic and progressive disease leads to an inevitable loss of autonomy (muscle weakness, respiratory and cardiac failure). With better multidisciplinary care, life expectancy has increased but also morbidity. From now one, the evaluation of the quality of life of children with DMD is necessary in therapeutic trials.

Given the specificities of the disease, it seems appropriate to have a specific scale. In the literature there isn't quality of life scale specific to Duchenne Muscular Dystrophy in French version. The only specific scale that exists is the specific module PedsQLTM DMD that was validated in English version in 2012. This scale is relevant for assessing the quality of life in clinical trials and in daily clinical practice given its psychometric properties (good internal consistency close to 0.8).The main hypothesis that we formulate is to validate the French translation of the pediatric module of Duchenne Muscular Dystrophy of the PedsQL ™ 3.0 scale.

ELIGIBILITY:
Inclusion Criteria:

* Boys aged 7 to 18, with genomic Duchenne muscular dystrophy whose parents (mother and / or father) or direct grandparents do not oppose.

Exclusion Criteria:

* Inability for the child to understand the issues
* Absence of direct parents or grandparents
* Child receiving antidepressant treatment
* Non French speaking child
* Duchenne Muscular Dystrophy girls

Ages: 5 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 105 boys with DMD distributed as follows: 35 patients with Duchenne muscular dystrophy by age category, 8-12 years old and 13-18 years old.
  For the 5-7 age group, only parents answer the questionnaire but medical data are collected.
  105 parents of boys with DMD, broken down as follows: 35 by age group (5-7, 8-12, 13-18)
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2018-09-19 (Actual); Primary Completion 2019-09-19 (Estimated); Study Completion 2019-09-19 (Estimated)

PRIMARY OUTCOMES:
Evaluate the validity of the French version of the DMD module of the PedsQLTM 3.0 scale | 12 months
  The validation process is confirmatory, the scale being widely used in English 201/5000 The internal consistency of the 4 dimensions of the PedsQL ™ DMD module will be evaluated by measuring the Cronbach Alpha. In terms of data availability to children (activity report).
  the validation of the DMD module will focus on the validity of constructs, internal structure validity, discriminant validity and reliability
Evaluate the reliability of the French version of the DMD module of the PedsQLTM 3.0 scale | 12 months
  PedsQLTM is a model for measuring quality of life in children with acute or chronic pathology. Pathology-specific PedsQL ™ provides a better assessment of the quality of life of this population

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Wallach, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No